CLINICAL TRIAL: NCT00264160
Title: Efficacy and Safety of Oral AMN107 in Adults With Chronic Myelogenous Leukemia Resistant and/or Intolerant to Imatinib Mesylate Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AIL01
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2012-08

CONDITIONS: Leukemia, Myeloid, Chronic
Keywords: AMN107; CML; Bcr Abl; cytogenetic response; Chronic Myelogenous Leukemia (CML); imatinib mesylate
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

ARMS (1):
- AMN107 (Experimental)
  Interventions: Drug: AMN107

INTERVENTIONS:
Drug: AMN107

SUMMARY:
This open-label, multicenter trial will evaluate the efficacy and safety of treatment with AMN107 in chronic myelogenous leukemia (CML) patients that are resistant and/or intolerant to imatinib mesylate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Imatinib - resistant or - intolerant Philadelphia chromosome-positive CML in blast crisis, accelerated or chronic phase
* Males or females ≥ 18 years of age

Exclusion Criteria:

* Impaired cardiac function
* Acute or chronic liver or renal disease
* Use of therapeutic coumadin
* Central nervous system (CNS) infiltration

Additional protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-05; Primary Completion 2008-11 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Cytogenetic response within 12 months | Every 6 months for 12 months

SECONDARY OUTCOMES:
To determine the rate of hematologic response at 12 months | Every Visit for 12 months
To determine the rate of molecular response at 12 months | Every 3 months for 12 months
To evaluate the time to cytogenetic and molecular response | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Litwinsky

REFERENCES:
- [Result] Kantarjian HM, Giles F, Gattermann N, Bhalla K, Alimena G, Palandri F, Ossenkoppele GJ, Nicolini FE, O'Brien SG, Litzow M, Bhatia R, Cervantes F, Haque A, Shou Y, Resta DJ, Weitzman A, Hochhaus A, le Coutre P. Nilotinib (formerly AMN107), a highly selective BCR-ABL tyrosine kinase inhibitor, is effective in patients with Philadelphia chromosome-positive chronic myelogenous leukemia in chronic phase following imatinib resistance and intolerance. Blood. 2007 Nov 15;110(10):3540-6. doi: 10.1182/blood-2007-03-080689. Epub 2007 Aug 22. PMID 17715389